CLINICAL TRIAL: NCT02548676
Title: Optical Angiography in Glaucoma
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Other Study IDs: OPHT - 110414
Record Dates: First submitted 2015-09-04; First posted 2015-09-14 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Glaucoma Patients: Patients with primary open angle glaucoma
  Interventions: Device: Optical angiography based on OCT
- Healthy controls: age- and sex matched controls
  Interventions: Device: Optical angiography based on OCT

INTERVENTIONS:
Device: Optical angiography based on OCT — This measurement will be obtained after the dilation of the pupil. Optical coherence tomography (OCT) is a non-invasive optical imaging modality enabling cross-sectional tomographic in vivo visualization of internal microstructure in biological systems. In ophthalmology OCT has become a standard device in visualizing the retina and is also considered a standard tool in the diagnosis of retinal disease. In optical angiography blood vessels contrasting against static tissue are visualized in a full depth resolved and label-free manner.

SUMMARY:
Glaucoma is one of the leading causes for blindness in industrialized countries. It is characterized by a progressive loss of retinal ganglion cells, morphological changes in the optic nerve head and a characteristic loss of visual field. It has been speculated for a long time that vascular factors may also contribute to the pathogenesis of the disease. This concept has been supported by several epidemiological studies showing that small retinal vessel calibre are associated with the disease. In the recent years tremendous enhancements in the field of optical coherence tomography has been achieved. These developments made it possible to visualize the retinal vasculature in a full depth manner without the application of an intravenous marker. The proposed study tests the hypothesis that patients with glaucoma show altered vascular morphology compared to healthy subjects. This is of importance because it may clarify the degree of vascular involvement in glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of manifest open angle glaucoma as defined as pathological optic disc appearance, glaucoma hemifield test outside normal limits and/or untreated IOP ≥ 21 mmHg on at least three measurements in the medical history. Mean deviation in the visual field test < 10dB

Exclusion Criteria:

* Normal ophthalmic findings, IOP ≤ 20mmHg
* No history of elevated IOP
* No signs of glaucomatous disc damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 open angle glaucoma patients 30 healthy age- and sex matched controls
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11-25 (Actual)

PRIMARY OUTCOMES:
Retinal vessel diameter as extracted from the angiograms | during the four weeks after the first screening day

SECONDARY OUTCOMES:
Systemic hemodynamics (Blood pressure) | during the four weeks after the first screening day
Intraocular pressure | during the four weeks after the first screening day
pulse | during the four weeks after the first screening day

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria